CLINICAL TRIAL: NCT05910853
Title: Whole Blood Biospecimen Collection for Subjects With Fanconi Anemia
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit new subjects due to disease rarity
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-09686
Record Dates: First submitted 2023-06-08; First posted 2023-06-20 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Fanconi Anemia (Non-Specific Genotypes): Cohort 1-Fanconi Anemia (Non-Specific Genotypes) (N=4):
  Inclusion:
  1. The participant is willing and able to provide written informed consent
  2. The participant is willing and able to provide appropriate photo identification
  3. Participants aged 18 to 85
  4. Participants have been diagnosed with Fanconi Anemia complementation group A*Inclusion preference (not required for enrollment into the study): 1)
  Participants preferentially have one of the following genotypes:
  c3788_3790delTCT, c295 G to T, c3558-3559 insertion of G, or c1115_1118delTTGG
  Exclusion:
  1. Participants who are pregnant or are nursing
  2. Participants with a known history of HIV, hepatitis, or other infectious diseases
  3. Participants who have taken an investigational product in the last 30 days Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
  Interventions: Diagnostic Test: Specimen Donation
- Fanconi Anemia (c3788_3790delTCT): Cohort 2 - Fanconi Anemia (c3788_3790delTCT) (N=1):
  Inclusion:
  1. The participant is willing and able to provide written informed consent
  2. The participant is willing and able to provide appropriate photo identification
  3. Participants aged 18 to 85
  4. Participants have been diagnosed with Fanconi Anemia complementation group A
  5. 1 participant must be diagnosed with the following genotype: c3788_3790delTCT
  Exclusion:
  1. Participants who are pregnant or are nursing
  2. Participants with a known history of HIV, hepatitis, or other infectious diseases
  3. Participants who have taken an investigational product in the last 30 days Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
  Interventions: Diagnostic Test: Specimen Donation
- Fanconi Anemia (c295 G to T): Cohort 3 - Fanconi Anemia (c295 G to T) (N=1):
  Inclusion:
  1. The participant is willing and able to provide written informed consent
  2. The participant is willing and able to provide appropriate photo identification
  3. Participants aged 18 to 85
  4. Participants have been diagnosed with Fanconi Anemia complementation group A
  5. 1 participant must be diagnosed with the following genotype: c295 G to T
  Exclusion:
  1. Participants who are pregnant or are nursing
  2. Participants with a known history of HIV, hepatitis, or other infectious diseases
  3. Participants who have taken an investigational product in the last 30 days Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
  Interventions: Diagnostic Test: Specimen Donation
- Fanconi Anemia (c3558-3559 insertion of G): Cohort 4 - Fanconi Anemia (c3558-3559 insertion of G) (N=1):
  Inclusion:
  1. The participant is willing and able to provide written informed consent
  2. The participant is willing and able to provide appropriate photo identification
  3. Participants aged 18 to 85
  4. Participants have been diagnosed with Fanconi Anemia complementation group A
  5. 1 participant must be diagnosed with the following genotype: c3558-3559 insertion of G
  Exclusion:
  1. Participants who are pregnant or are nursing
  2. Participants with a known history of HIV, hepatitis, or other infectious diseases
  3. Participants who have taken an investigational product in the last 30 days Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
  Interventions: Diagnostic Test: Specimen Donation
- Fanconi Anemia (c1115_1118delTTGG): Cohort 5 - Fanconi Anemia (c1115_1118delTTGG) (N=1):
  Inclusion:
  1. The participant is willing and able to provide written informed consent
  2. The participant is willing and able to provide appropriate photo identification
  3. Participants aged 18 to 85
  4. Participants have been diagnosed with Fanconi Anemia complementation group A
  5. 1 participant must be diagnosed with the following genotype: c1115_1118delTTGG
  Exclusion:
  1. Participants who are pregnant or are nursing
  2. Participants with a known history of HIV, hepatitis, or other infectious diseases
  3. Participants who have taken an investigational product in the last 30 days Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
  Interventions: Diagnostic Test: Specimen Donation

INTERVENTIONS:
Diagnostic Test: Specimen Donation — Blood donation

SUMMARY:
The primary study objective is to collect biospecimen samples (e.g., blood) from participants diagnosed with Fanconi Anemia. The biospecimens will be used to create a biorepository that can be used to identify disease associated biomarkers and potential targets with immune and multi-omics profiling. The disease sample collection and analysis will be the foundation for an extensive network of biospecimen access and linked datasets for future translational research.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to provide written informed consent
* The participant is willing and able to provide appropriate photo identification
* Participants aged 18 to 85
* Participants have been diagnosed with Fanconi Anemia complementation group A

Exclusion Criteria:

* Participants who are pregnant or are nursing
* Participants with a known history of HIV, hepatitis, or other infectious diseases Participants who have taken an investigational product in the last 30 days Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have been diagnosed with Fanconi Anemia
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Biospecimen Samples collect from patients with Fanconi Anemia participants diagnosed with Fanconi Anemia. | 1 year
  The primary study objective is to collect biospecimen samples (e.g., blood) from participants diagnosed with Fanconi Anemia. The biospecimens will be used to create a biorepository that can be used to identify disease associated biomarkers and potential targets with immune and multi-omics profiling. The disease sample collection and analysis will be the foundation for an extensive network of biospecimen access and linked datasets for future translational research.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Frisina, M.S., Study Chair — Sanguine Biosciences
Locations (1):
- Sanguine Biosciences, Woburn, Massachusetts, United States